CLINICAL TRIAL: NCT03675022
Title: Effect of Dupilumab on Sleep Apnea Severity in Patients With Chronic Rhinosinusitis
Brief Title: Effect of Dupilumab on Sleep Apnea in Patients With Rhinosinusitis
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Inability to recruit during COVID
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Tanya Laidlaw, MD, Director of Translational Research in Allergy, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P001031
Record Dates: First submitted 2018-07-18; First posted 2018-09-18 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Sleep Apnea; Rhinosinusitis Chronic
MeSH Terms: conditions — Sleep Apnea Syndromes | interventions — dupilumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dupilumab (Experimental): Dupilumab injections every 2 weeks.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — The investigational drug is dupilumab, 300mg in 2ml solution for subcutaneous application. All Patients will receive dupilumab, 300mg, every two weeks (8 subcutaneous injections total).
  Other Names: Dupixent

SUMMARY:
Obstructive Sleep Apnea (OSA) is a common disorder with serious consequences that remains underrecognized, with >80% of OSA patients undiagnosed, and undertreated due to inadequate treatment options. The development of additional treatments for OSA, such as pharmacotherapy, are critically needed.

The collaboration between Regeneron and Sanofi are funding this project. Regeneron will be providing the drug and the contract will be with Regeneron. Both companies are involved as it is a collaboration across the companies.

DETAILED DESCRIPTION:
Clinical Background on OSA OSA is a prevalent disorder, with roughly 1 in 5 adults estimated to have at least mild OSA and 1 in 15 estimated to have at least moderate OSA. Furthermore, OSA causes a number of adverse cardiovascular, neurocognitive, and daytime functional consequences. As a result, understanding the pathophysiology and developing treatments is a major public health goal. Unfortunately, only approximately 50% of patients tolerate the main therapy for OSA, Continuous Positive Airway Pressure (CPAP). Therefore, new therapeutic approaches are clearly needed.

OSA is caused by collapse of the pharyngeal airway during sleep due to the sleep state-related loss of pharyngeal muscle activity. High nasal resistance can contribute to pharyngeal collapse as well by increasing the suction pressure downstream in the velo- and oropharynx. In fact, a recent study in 139 patients with chronic rhinosinusitis (CRS) demonstrated an extremely high prevalence of OSA (65% of the CRS patients had OSA compared to a prevalence in the normal population of 5-15%). Therefore, a drug that reduces nasal congestion and pharyngeal edema, such as dupilumab, could potentially improve OSA in some patients.

Immunologic Background on OSA and role of Type 2 inflammation Indeed, preliminary patient-reported outcomes data from early clinical trials with dupilumab have shown that dupilumab treatment of patients with sinus disease reduces reports of nocturnal awakenings, as well as sleep-related outcomes on the SinoNasal Outcome Test (SNOT-22). In addition to the known effects of dupilumab on the reduction of nasal polyp size/volume, there is ample evidence to propose that the specific anti-inflammatory effects achieved with IL-4Rα blockade will be particularly relevant to a potential therapeutic effect of dupilumab on OSA in patients with comorbid CRS. There are a number of Type 2 inflammatory markers that are increased in patients with CRS and OSA, which taken together suggest that OSA in these patients is truly an inflammatory disease, and not solely a disease of abnormal anatomy. Serum IL-4 levels are elevated in patients with rhinitis and OSA, and those levels are negatively correlated with time spent in REM sleep. Furthermore, two inflammatory markers of mast cell activation, urinary leukotriene E4 and urinary prostaglandin D2, are also known to be elevated in OSA, likely due to the increased chronic mast cell stimulation afforded by the high circulating IL-4 levels. Strikingly, both urinary leukotriene E4 and prostaglandin D2 levels correlate with OSA severity, as measured by either percentage of overnight time spent with SaO2 <90% or the apnea/hypopnea index (AHI).

There is additional clinical evidence to suggest that OSA may be more than "just" an anatomic disease. Although endoscopic sinus surgery to remove inflamed sinus tissue in patients with OSA and CRS does improve OSA symptoms, non-surgical anti-inflammatory treatments, including intranasal steroids and leukotriene modification with montelukast, have also been found to improve OSA symptoms and decrease the AHI.

Given these immunological findings, the investigators suspect that extensive Type 2 inflammation is a major contributing factor for patients with CRS and OSA, and that IL-4Rα blockade will be a powerful therapeutic tool in sleep apnea. In combination with the preliminary patient-reported outcomes data suggesting that dupilumab improves sleep quality, the investigators feel confident that dupilumab will successfully provide a clinically-quantifiable therapeutic improvement on the severity of OSA in patients with CRS and OSA. As there are currently no FDA-approved medications for the treatment of OSA, and 65% of all patients with CRS suffer from OSA, the investigators feel as though positive results from this pilot trial would be a powerful step towards providing a new biologic therapy to an underserved medical population.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 to 65 years)
* BMI < 35 kg/m2
* Bilateral CRS (clinical diagnosis) with or without nasal polyposis despite intranasal corticosteroid treatment for at least 3 months.
* Patients will be required to report at least 2 of the following symptoms prior to screening: (1) nasal obstruction/blockage, (2) nasal discharge or discolored postnasal drainage, (3) facial pain or pressure, and (4) reduction or loss of sense of smell, with symptom duration of at least 3 months.
* Suffering from OSA with AHI > 10 episodes/hr based on the home sleep test (described below) and not using CPAP.
* Willing, committed, and able to return for all clinic visits and complete all study-related procedures.
* In females of childbearing potential: Negative pregnancy test. A urine pregnancy test will be performed in each site visit to ensure that the patients are not pregnant while using dupilumab.

Exclusion Criteria:

* Concurrent sleep disorder
* Previous participation in any clinical trial of dupilumab in which active treatment was administered.
* Oral corticosteroids, monoclonal antibodies, immunosuppressive treatment, or anti-immunoglobulin E (anti-IgE) therapy during the 6 weeks preceding the screening.
* Concomitant conditions making them not evaluable for the primary endpoint. Prior diagnosis of OSA will not be exclusionary.
* Lactating females or pregnant females.
* Subjects for whom there is concern about compliance with the protocol procedures.
* Any medical condition which, in the opinion of the Investigator, would interfere with participation in the study or place the subject at risk (chronic infectious diseases such as TB, HIV, Hepatitis, etc.).
* History of hypersensitivity to the study drug.
* History of substance abuse (drug or alcohol) or any other factor (e.g., serious psychiatric condition) that could limit the subject's ability to comply with study procedures.
* Subjects must refrain from intranasal decongestants for 1 week prior to starting the study.
* Subjects with a medical history of HSV1 or HSV2, or with a history of recurrent conjunctivitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Percent change in apnea-hypopnea index (AHI) after 16 weeks of dupilumab therapy | 16 weeks
  The effect of dupilumab on OSA severity in patients with nasal obstruction due to chronic rhinosinusitis with or without nasal polyposis (Bilateral CRS). AHI is the amount of respiratory events that a patient has per hours of sleep.

SECONDARY OUTCOMES:
Effect of 16 weeks of dupilumab on sleep architecture total sleep time | 16 weeks
  Sleep architecture variables as measured with in-laboratory sleep study of total sleep time
Effect of 16 weeks of dupilumab on sleep architecture sleep stage percentages | 16 weeks
  Sleep architecture variables as measured with in-laboratory sleep study of sleep stage percentages
Effect of 16 weeks of dupilumab on sleep architecture arousal index | 16 weeks
  Sleep architecture variables as measured with in-laboratory sleep study of arousal index. The arousal index is how many times a subject wakes up per hour during sleep.
Effect of 16 weeks of dupilumab on sleep architecture oxygen saturation | 16 weeks
  Sleep architecture variables as measured with in-laboratory sleep study of oxygen saturation
Epworth Sleepiness Score (ESS) | 16 weeks
  Epworth Sleepiness Score (ESS) - The ESS asks the respondent to rate on a 4-point scale (0-3) their usual chances of having dozed off or fallen asleep while engaged in eight different activities that differ widely in their somnificity. The total ESS score (the sum of 8 item-scores) gives an estimate of a more general characteristic, the person's 'average sleep propensity' or ASP, across a wide range of activities in their daily lives. Scores range from 0 to 24, 0 being not sleepy at all and 24 being the most sleepy.
Pittsburgh Sleep Quality Index (PSQI) | 16 weeks
  Pittsburgh Sleep Quality Index (PSQI) - The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month. A total score of "5" or greater is indicative of poor sleep quality. If you scored "5" or more it is suggested that you discuss your sleep habits with a healthcare provider. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality. A higher score indicates that a person generally has difficulty carrying out certain activities because you are too sleepy or tired.
Functional Outcomes of Sleep Quality (FOSQ) | 16 weeks
  Functional Outcomes of Sleep Quality (FOSQ) - Disease specific quality of life questionnaire to determine functional status in adults; measures are designed to assess the impact of disorders of excessive sleepiness on multiple activities of everyday living and the extent to which these abilities are improved by effective treatment. This scale has 30 items, 5 factor subscales, scaling of items is 0-4. To obtain total score, take all the subscale scores and calculate the mean of these scores and then multiply that mean by five. The potential range of scores for the total score is 5-20.
Subjective sleep quality [visual analog scale(VAS)] | 16 weeks
  Subjective sleep quality [visual analog scale(VAS)] - on a scale of 1-10, subjects answer questions on how sleepy they are with 0 being least sleepy and 10 being most sleepy
Effect of 16 weeks of dupilumab on nasal resistance with catheter | 16 weeks
  Effect of 16 weeks of dupilumab on awake nasal resistance measurements using a pressure catheter
Effect of 16 weeks of dupilumab on nasal resistance with mask | 16 weeks
  Effect of 16 weeks of dupilumab on awake nasal resistance measurements using a mask with pneumotach

OTHER OUTCOMES:
Sino-Nasal Outcome Test (SNOT-22) | 16 weeks
  Effect of 16 weeks of dupilumab on the 22 item Sino-Nasal Outcome Test (SNOT-22)
Visual analog scale (VAS) for rhinosinusitis | 16 weeks
  Effect of 16 weeks of dupilumab on the Visual analog scale (VAS) for rhinosinusitis. - on a scale of 1-10, subjects answer questions on their rhinosinusitis symptom with 0 being least severe and 10 being most severe
University of Pennsylvania Smell Identification Test (UPSIT) | 16 weeks
  Effect of 16 weeks of dupilumab on smell identification, using the University of Pennsylvania Smell Identification Test (UPSIT)
Effect of 16 weeks of dupilumab on peak nasal inspiratory flow (PNIF) | 16 weeks
  Effect of 16 weeks of dupilumab on peak nasal inspiratory flow (PNIF)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States